CLINICAL TRIAL: NCT04646239
Title: Determining Biomarkers of Trained Immunity in a Randomized Controlled Trial of the Measles, Mumps, and Rubella Vaccine - a Sub-study of the CROWN CORONATION Trial
Brief Title: Biomarkers of Trained Immunity Following MMR Vaccination
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Michael Avidan, Professor, Washington University School of Medicine
Other Study IDs: 202011081
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: COVID 19; Trained Immunity; Infectious Diseases
MeSH Terms: conditions — COVID-19; Communicable Diseases | interventions — DNA Mismatch Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 45 mL peripheral blood drawn around 60 to 90 days after last SARS-CoV-2 vaccine injection. De-identified plasma and peripheral blood mononuclear cells will be extracted from the collected specimens and stored for analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants in the CROWN CORONATION trial: The CROWN CORONATION trial will randomly allocate adult participants to a single intramuscular injection of MMR vaccine or Placebo (0.9% saline). All participants in this sub-study receive SARS-CoV-2 specific vaccine subsequent to the MMR or Placebo injection.
  Interventions: Diagnostic Test: Heterologous stimuli; Diagnostic Test: Neutralization assay

INTERVENTIONS:
Diagnostic Test: Heterologous stimuli — In vitro exposure of peripheral blood mononuclear cells to heterologous stimuli
  Other Names: For example; RPMI medium, MMR, SARS-CoV-2, Influenza, TLR3 ligand, TLR7/8 ligand, TLR4 ligand
Diagnostic Test: Neutralization assay — In vitro measurement of neutralizing antibody activity to wild-type SARS-CoV-2

SUMMARY:
This is a substudy of NCT04333732. The goal of this sub-study is to identify and characterize biomarkers of trained immunity by measuring, in vitro, immune responses to heterologous products, especially viral associated products, in the MMR vaccinated compared placebo groups.

All participants are randomly assigned to MMR or placebo injection at baseline, followed by SARS-CoV-2 specific vaccination. Blood is drawn around 60 to 90 days after the last SARS-CoV-2 specific vaccine injection.

DETAILED DESCRIPTION:
A sub-study of the CROWN CORONATION Trial (COVID-19 Research Outcomes Worldwide Network for CORONAvirus prevenTION; NCT04333732). The goal of this sub-study is to identify and characterize biomarkers of trained immunity by measuring, in vitro, immune responses to heterologous products, especially virally associated products, in those exposed to MMR vaccine injection compared to those exposed to 0.9% sodium chloride ('normal saline') placebo injection.

A secondary objective is comparison of SARS-CoV-2 neutralization assays between MMR and placebo comparison groups around 60 to 90 days after the last SARS-CoV-2 specific vaccine injection.

All participants are randomly assigned to MMR or placebo injection at baseline, followed by SARS-CoV-2 specific vaccination. Blood is drawn around 60 to 90 days after the last SARS-CoV-2 specific vaccine injection. Peripheral blood mononuclear cells (PMBC) will be isolated from samples and stimulated with heterologous products (for example; Roswell Park Memorial Institute medium [RPMI; negative control], MMR [the vaccine itself as specific stimulus], severe acute respiratory syndrome coronavirus-2 [SARS-CoV-2; heat inactivated], influenza virus [heat inactivated], toll-like receptor 3 ligand [TLR3 ligand; poly I:C], toll-like receptor 7/8 ligand [TLR7/8 ligand; R848], toll-like receptor 4 ligand [TLR4 ligand; lipopolysaccharide (LPS)]). Supernatants will be assayed by multiplex luminex protein assay at 24 hr (for example; type I interferons [IFN], interleukin [IL]-1β , IL-6, tumor necrosis factor [TNF]-α) and after 5 days (for example; IFN-γ, IL-17, IL-22, IL-10). This process of testing stimulus-response will be conducted on both the baseline and day 30 samples, collected from both the MMR and Placebo groups.

Neutralization assay will be conducted on all samples using wild-type SARS-CoV-2.

Measles IgG titres will be measured on all samples. Measles IgG titres will be used for sensitivity analysis.

ELIGIBILITY:
Inclusion/ Exclusion Criteria:

Prospective participant must already be enrolled into the CROWN CORONATION trial at the sub-study location. Refer to NCT04333732 for list of inclusion / exclusion criteria for the study population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The CROWN CORONATION trial enrolls adults at risk of developing COVID-19 due to their work in the healthcare environment. To be eligible, prospective participants for the CROWN CORONATION trial must not have a contra-indication to receiving the live attenuated Measles, Mumps and Rubella vaccine (MMR) and must not be exposed to agents that may complicate the interpretation of findings regarding the hypothesized protective effect of MMR for the prevention of COVID-19. The sub-study will consecutively approach all participants enrolled in the CROWN CORONATION trial to elicit enrolment in the sub-study cohort.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Cytokine (or chemokine) production in response to heterologous stimuli | Around 60 to 90 days after last SARS-CoV-2 specific vaccine injection
  Cytokines such as TNF-α, IL-1β and IL-6 produced by human monocytes, and IFN-γ produced by natural killer (NK)-cells, are markers of trained immunity and these (and other cytokines and chemokines) will be measured in supernatants of stimulated PBMCs from a cohort of participants in the CROWN CORONATION trial. All cytokines and chemokines are measured in picograms/milliliter.

SECONDARY OUTCOMES:
Neutralization assay | Around 60 to 90 days after last SARS-CoV-2 specific vaccine injection
  Neutralizing antibody activity to wild-type SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Avidan, MD, Principal Investigator — Washington Univeristy School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The project team will make the de-identified data available to the public within 1 year after publication using a public repository. Prior to that time, data will be deposited in the Washington University Open Scholarship repository. Any request for data not deposited in the repository must be directed to the Principal Investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 Year

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT04646239/SAP_000.pdf